CLINICAL TRIAL: NCT03311386
Title: Evaluation of Collateral Vessels in Patients With Acute Ischemic Stroke Receiving Thrombolytic Therapy (Clinical and Radiological Study)
Brief Title: Intracranial Collaterals in Acute Stroke and Clinical Outcome
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mamdouh Mohammed Tawfeeq, principle investigator, Assiut University
Other Study IDs: Collaterals and acute stroke
Record Dates: First submitted 2017-10-02; First posted 2017-10-17 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Collateral Circulation, Any Site
MeSH Terms: interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in AIS receiving actilyse: the patients will receive actilyse intaravenously in a dose of 0.9mg/kg once
  Interventions: Drug: Actilyse

INTERVENTIONS:
Drug: Actilyse — thrombolytic therapy
  Other Names: Alteplase

SUMMARY:
Assessment of the evolution of intracranial collaterals and its relationship with functional outcomes in acute ischemic stroke (AIS) patients treated with IV tissue plasminogen activator (tPA).

DETAILED DESCRIPTION:
Intracranial collaterals Assessment in acute ischemic stroke In clinical practice, infarct growth does not always progress to involve the full extent of the vascular territory, even if the affected intracranial artery fails to recanalize. The presence and recruitment of various collateral channels are believed to be responsible for this phenomenon in acute ischemic stroke (AIS). These collaterals may also play an important role in influencing the safety and efficacy of acute revascularization approaches. Although blood supply from the leptomeningeal collaterals may temporarily maintain the ischemic penumbra, the persistence and effectiveness of this alternative circulatory supply is erratic and unpredictable. Some collaterals may disappear over time (collateral failure); this is one of the mechanisms responsible for clinical deterioration following initial improvement.

Conversely, dramatic resolution of initial neurologic deficits may be seen though the occluded intracranial artery did not recanalize, often attributable to the rapid improvement of cerebral perfusion via effective collateral pathways (collateral recruitment). Therefore, the temporal behavior of intracranial collaterals may play an important role in determining the functional outcome in AIS patients.

CT angiography (CTA) of the brain is acutely performed in AIS patients before or immediately after administering IV tissue plasminogen activator (tPA) The Alberta Stroke Program Early CT (ASPECTS) leptomeningeal collaterals score on CT-angiography helps in prognosticating functional outcome in acute ischemic stroke (AIS) patients treated with intravenous thrombolysis. Leptomeningeal collaterals in AIS are dynamic, especially during the first few hours or days of AIS.

In animals, 3 different types of collaterals have been identified: transient collaterals that could be seen immediately after the stroke and last less than 90 minutes; impermanent collaterals that disappear after 90-150 minutes; and persistent collaterals, which can be seen for longer periods.

Patients with good collateral flow demonstrated less hypo perfused tissue and less infarct growth within the penumbra zone than those with poor collateral . A relationship is found between good early collaterals on pretreatment imaging and smaller infarct volume with better outcomes.

The initial state of the collateral circulation on the pretreatment CTA also has bearing on the clinical effect of the collateral recruitment on the day 2 CTA.

However, collateral recruitment with poor pretreatment collaterals was associated with poor functional outcome at 3 months and a higher risk of intracranial hemorrhage.

One plausible mechanism that delayed collateral recruitment lead to worse outcomes could be related to the maximal vasodilation in the ischemic area and how collateral recruitment in the adjacent regions may trigger a steal-like phenomenon with resultant expansion of the ischemic core. Another possible mechanism could be related to failed autoregulation in the affected vascular territory, leading to increased hyper perfusion damage with a higher chance of bleeding.

ELIGIBILITY:
IInclusion Criteria:

* Patient presenting to the emergency department with symptoms consistent with ischemic stroke.
* Age > 18 yrs.
* Evidence of a visible and symptomatic intracranial occlusion on baseline CT-angiography (intracranial ICA, M1 MCA segment +/- intracranial ICA, proximal M2 MCA).
* Treatment with IV tPA.

Exclusion Criteria:

* Intracranial hemorrhage (ICH) identified on baseline CT.
* Previous moderate to large stroke in the ipsilesional hemisphere.
* Modified Rankin Scale > 2 at baseline.
* Unable to have CT-angio performed due to recent estimated creatinine clearance eCCr<60 ml/min, contrast allergy or other reasons.
* Any terminal illness (patient not expected to survive > 1 year).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute ischemic stroke within 4.5 hours - legible for receiving IV r TPA- admitted to Neurology department of Asyut University within 1 year (2017-2018)
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
90-days functional outcome | 90 days
  90-day modified Rankin Score (mRS) 0-2 or equal to the pre-stroke modified Rankin scale he Modified Rankin Scale (mRS) The scale runs from 0-6 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

SECONDARY OUTCOMES:
Early neurologic improvement | 24 hours
  Defined as The National Institutes of Health Stroke Scale score "NIHSS" of 0 to 2 at 24 hours or an 8-point drop in NIHSS score from baseline to 24 hours.
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, 0 No stroke symptoms 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke

CONTACTS AND LOCATIONS:
Overall Officials: Essam Darwish, Professor, Principal Investigator — Assiut University; Ahmed Hamdy, Ass.Prof, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Bang OY, Goyal M, Liebeskind DS. Collateral Circulation in Ischemic Stroke: Assessment Tools and Therapeutic Strategies. Stroke. 2015 Nov;46(11):3302-9. doi: 10.1161/STROKEAHA.115.010508. Epub 2015 Oct 8. No abstract available. PMID 26451027